CLINICAL TRIAL: NCT01697254
Title: The CARRA Registry
Acronym: CARRA Registry
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH); Arthritis Foundation (Other); Lupus Foundation of America (Other); Cure JM Foundation (Unknown)
Responsible Party: Sponsor
Other Study IDs: Pro00018979; 1RC2AE058934-01
Record Dates: First submitted 2012-09-28; First posted 2012-10-02 (Estimated); Last update posted 2015-11-17 (Estimated); Status verified 2015-11

CONDITIONS: Juvenile Idiopathic Arthritis; Systemic Lupus Erythematosus; Mixed Connective Tissue Disease; Juvenile Ankylosing Spondylitis; Juvenile Dermatomyositis; Localized Scleroderma; Systemic Sclerosis; Vasculitis; Sarcoid; Fibromyalgia, Primary; Auto-inflammatory Disease; Idiopathic Uveitis Idiopathic
MeSH Terms: conditions — Arthritis, Juvenile; Lupus Erythematosus, Systemic; Mixed Connective Tissue Disease; Dermatomyositis; Scleroderma, Localized; Scleroderma, Systemic; Vasculitis; Sarcoidosis; Fibromyalgia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — Specimens currently being collected from subjects with juvenile dermatomyositis JDM), systemic juvenile idiopathic arthritis (sJIA), and localized scleroderma.
Oversight: Data Monitoring Committee: No

SUMMARY:
This CARRA Registry study will create a foundational database for rheumatic diseases of childhood using a novel informatics infrastructure developed as part of the larger clinical project. The creation of a CARRA-wide informatics infrastructure will enable efficient, observational, disease-related data capture across all CARRA sites for pediatric rheumatic diseases. The CARRA Registry study will demonstrate the feasibility of expanding to more data intensive registries for observational studies, comparative effectiveness research, pharmaceutical clinical trials and translational research.

DETAILED DESCRIPTION:
This protocol represents one aim of a larger clinical project that will advance the infrastructure of the Childhood Arthritis and Rheumatology Research Alliance (CARRA) network, facilitate expanded clinical and translational pediatric research, and rapidly transform the culture of pediatric rheumatology toward universal participation in research. Through the creation of sophisticated informatics infrastructure, provision of comprehensive site support and the engagement of families, patients, and communities, CARRA will provide the opportunity for affected children at every CARRA site to participate in high quality clinical and translational research.

The larger clinical project includes development of a CARRA-wide informatics platform with capabilities for capture, storage, visualization, and secure HIPAA-compliant sharing of validated disease metrics and relevant subject demographics, utilizing centralized Electronic Data Capture (EDC) and phone interviews where appropriate, and ontology-based data storage using a distributed database structure based on the NIH-supported i2b2 (Informatics Integrating Biology and the Bedside) framework. This will enable efficient, observational, disease-related data capture across CARRA sites. The CARRA Registry described in this protocol will form the foundational database and will involve the capture of data including pediatric rheumatic diseases as described in Appendix A.

The CARRA Registry will support data collection from the use of consensus treatment plans (CTPs), clinical trials, observational disease registries, comparative effectiveness research, and other research on patients with pediatric rheumatic disease. The CARRA Registry will form the basis for future CARRA studies and the Duke Clinical Research Institute (DCRI) is serving as the CARRA Data Coordinating Center (DCC) for this protocol.

ELIGIBILITY:
Inclusion Criteria:

* Onset of rheumatic disease prior to age 16 years for JIA and onset prior to age 18 years for all other rheumatic diseases
* Subject has been diagnosed with a defined pediatric rheumatic disease including: Mixed Connective Tissue Disease (MCTD), Systemic Lupus Erythematosus (SLE), Primary Sjögren's Syndrome (pSS), Systemic Sclerosis (SS), Juvenile Dermatomyositis (JDM), Localized Scleroderma (LS), Juvenile Idiopathic Arthritis (JIA), Vasculitis, Sarcoid, Auto-inflammatory Diseases, Idiopathic Uveitis (IU), and Juvenile Primary Fibromyalgia Syndrome (JPFS).
* Subject (and/or parent/legal guardian when required) is able to provide written informed consent and willing to comply with study procedures.

Exclusion Criteria:

- None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects will be recruited from the patient population of a CARRA Registry site.
Sampling Method: Non-Probability Sample
Enrollment: 9587 (Actual)
Dates: Start 2009-08; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Enrolled Subjects | baseline
  This is an observational registry. The primary outcome is the # of subjects enrolled with pediatric rheumatic disease.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Schanberg, MD, Principal Investigator — Duke University; Norman T Illowite, MD, Principal Investigator — Children's Hospital at Montefiore; Christy Sandborg, MD, Principal Investigator — Lucile Salter Packard Children's Hospital/Stanford University School of Medicine; Carol Wallace, MD, Principal Investigator — Seattle Children's Hospital/ University of Washington School of Medicine
Locations (1):
- Duke Clinical Research Institute, Durham, North Carolina, United States

REFERENCES:
- [Background] Robinson AB, Hoeltzel MF, Wahezi DM, Becker ML, Kessler EA, Schmeling H, Carrasco R, Huber AM, Feldman BM, Reed AM; Juvenile Myositis CARRA Subgroup, for the CARRA Registry Investigators. Clinical characteristics of children with juvenile dermatomyositis: the Childhood Arthritis and Rheumatology Research Alliance Registry. Arthritis Care Res (Hoboken). 2014 Mar;66(3):404-10. doi: 10.1002/acr.22142. PMID 23983017
- [Result] Natter MD, Quan J, Ortiz DM, Bousvaros A, Ilowite NT, Inman CJ, Marsolo K, McMurry AJ, Sandborg CI, Schanberg LE, Wallace CA, Warren RW, Weber GM, Mandl KD. An i2b2-based, generalizable, open source, self-scaling chronic disease registry. J Am Med Inform Assoc. 2013 Jan 1;20(1):172-9. doi: 10.1136/amiajnl-2012-001042. Epub 2012 Jun 25. PMID 22733975
- [Result] Beukelman T, Ringold S, Davis TE, DeWitt EM, Pelajo CF, Weiss PF, Kimura Y; CARRA Registry Investigators. Disease-modifying antirheumatic drug use in the treatment of juvenile idiopathic arthritis: a cross-sectional analysis of the CARRA Registry. J Rheumatol. 2012 Sep;39(9):1867-74. doi: 10.3899/jrheum.120110. Epub 2012 Aug 1. PMID 22859354
- [Result] Ringold S, Beukelman T, Nigrovic PA, Kimura Y; CARRA Registry Site Principal Investigators. Race, ethnicity, and disease outcomes in juvenile idiopathic arthritis: a cross-sectional analysis of the Childhood Arthritis and Rheumatology Research Alliance (CARRA) Registry. J Rheumatol. 2013 Jun;40(6):936-42. doi: 10.3899/jrheum.121147. Epub 2013 Apr 15. PMID 23588937
- [Result] Weiss PF, Beukelman T, Schanberg LE, Kimura Y, Colbert RA; CARRA Registry Investigators. Enthesitis-related arthritis is associated with higher pain intensity and poorer health status in comparison with other categories of juvenile idiopathic arthritis: the Childhood Arthritis and Rheumatology Research Alliance Registry. J Rheumatol. 2012 Dec;39(12):2341-51. doi: 10.3899/jrheum.120642. Epub 2012 Oct 15. PMID 23070991
- [Result] Kimura Y, Weiss JE, Haroldson KL, Lee T, Punaro M, Oliveira S, Rabinovich E, Riebschleger M, Anton J, Blier PR, Gerloni V, Hazen MM, Kessler E, Onel K, Passo MH, Rennebohm RM, Wallace CA, Woo P, Wulffraat N; Childhood Arthritis Rheumatology Research Alliance Carra Net Investigators. Pulmonary hypertension and other potentially fatal pulmonary complications in systemic juvenile idiopathic arthritis. Arthritis Care Res (Hoboken). 2013 May;65(5):745-52. doi: 10.1002/acr.21889. PMID 23139240
- [Derived] Kimura Y, Grevich S, Beukelman T, Morgan E, Nigrovic PA, Mieszkalski K, Graham TB, Ibarra M, Ilowite N, Klein-Gitelman M, Onel K, Prahalad S, Punaro M, Ringold S, Toib D, Van Mater H, Weiss JE, Weiss PF, Schanberg LE; CARRA Registry Investigators. Pilot study comparing the Childhood Arthritis & Rheumatology Research Alliance (CARRA) systemic Juvenile Idiopathic Arthritis Consensus Treatment Plans. Pediatr Rheumatol Online J. 2017 Apr 11;15(1):23. doi: 10.1186/s12969-017-0157-1. PMID 28399931